CLINICAL TRIAL: NCT03270410
Title: Design of a Non-invasive Multi-modal Neonatal Monitoring System: Preliminary Observational Study
Brief Title: Design of a Non-invasive Multi-modal Neonatal Monitoring System
Acronym: VARI-NEONAT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3012
Record Dates: First submitted 2017-08-23; First posted 2017-09-01 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Neonatal Disorder
Keywords: neonates; non invasive monitoring
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates: Babies born in Rennes University Hospital
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — After parental information and collection of their non-opposition, the data of the daily cardio-respiratory recordings of the newborns hospitalized in the units of Neonatology are collected and analyzed.
  At the same time, a video recording is set up. This video recording does not modify the care provided for the child, the organization of the day with nursing and parental care.

SUMMARY:
This is a preliminary study whose objectives are to define the clinical use cases and the constraints of the implementation of a multi-sensor image-sound system.

DETAILED DESCRIPTION:
300 000 newborns per year are hospitalized in European neonatal units in the post-natal period. This is a critical period for neurobehavioral development and the establishment of an optimal model of sleep-wake cycle is fundamental for brain development.

The objective of the research is to develop new tools for computer-aided clinical and predictive diagnosis and real-time monitoring in neonatology.

The development of non-invasive sensors based on video and sound images aims to improve the short- and medium-term prognosis in perinatal patients.

To that aim, multi-modal composite indices integrating the image (which is used only to generate a quantification of the movement) and the sound to the bioelectric signals already available (electrocardiogram, oxymetry, temperature) will be developed to provide diagnostic and prognostic information.

ELIGIBILITY:
Inclusion Criteria:

* newborns less than 6 weeks old in corrected terms;
* newborns in one of the following situations:

  * persistent discomfort (apneas);
  * infection or suspicion of infection;
  * premature with uncomplicated evolution;
  * Premature brain lesion acquired in perinatal;
  * newborn having been exposed to premature rupture of the membranes.

Exclusion Criteria:

* Congenital malformation;
* Metabolic disease.

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is aimed at newborns hospitalized at the CHU in Rennes
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Evolution of the cardiac variability during the stay in the ward | Up to 2 months
  The cardiac signals collected by the clinical monitoring required for hospitalization in a neonatal unit will be analyzed by specific routines to calculate parameters of cardiac variability.

SECONDARY OUTCOMES:
Evolution of the respiratory variability during the stay in the ward | Up to 2 months
  The respiratory signals collected by the clinical monitoring required for hospitalization in a neonatal unit will be analyzed by specific routines to calculate parameters of respiratory variability.
Evolution of the babies' movements during the stay in the ward | Up to 2 months
  Continuous video acquisitions of the newborns are realized. Video images will be analyzed by specific routines to extract quantitative parameters of movements.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PLADYS, MD, PhD, Study Director — CHU Rennes
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No